CLINICAL TRIAL: NCT04340037
Title: A Pre-operative Nomogram for Sepsis After Percutaneous Nephrolithotomy Treating Solitary, Unilateral, and Proximal Ureteral Stones
Brief Title: Prediction of Sepsis After Percutaneous Nephrolithotomy
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Li Cong, Professor, Tongji Hospital
Other Study IDs: 2019S1035v2
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Percutaneous Nephrolithotomy; Infection; Urolithiasis; Albumin Globulin Ratio
MeSH Terms: conditions — Infections; Urolithiasis | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- proximal ureteral stone patient: Patients underwent percutaneous nephrolithotomy treating unilateral, solitary and proximal ureteral stones.
  Interventions: Procedure: percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: percutaneous nephrolithotomy — percutaneous surgery using nephroscope

SUMMARY:
We aim to determine the preoperative predictors of sepsis after percutaneous nephrolithotomy (PCNL) in patients with unilateral, solitary and proximal ureteral stones.

ELIGIBILITY:
Inclusion Criteria:

* (1) PCNL was performed to treat unilateral, solitary, and proximal ureteral stones; and (2) age ≥18 years

Exclusion Criteria:

* anatomical renal abnormalities (horseshoe kidney, solitary kidney, transplant kidney and kidney duplication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 745 patients who underwent PCNL from January 2012 to December 2018 were enrolled when meeting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 745 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
sepsis | within 48 hour after surgery
  the concurrence of infection and a minimum of two of the following within 48 hours of surgery: (1) heart rate >90/minute, (2) body temperature >38°C, (3) leukocyte count <4,000 cells/μL or >12,000 cells/μL, and (4) respiratory rate >20/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The data is not suitable to be public